CLINICAL TRIAL: NCT04236921
Title: A Phase 1 Study to Evaluate the Bioequivalence Between DopaSnap® (Carbidopa/Levodopa 25/100 mg Tablet) and Carbidopa/Levodopa 25/100 mg Tablet and to Evaluate the Food-Effect of DopaSnap® in Normal Healthy Volunteers
Brief Title: Bioequivalence Bewteen DopaSnap® (Cabidopa/Levopdoap 25/100 mg Tablet) and Carbidopa/Levodopa 25/100 mg Tablet (Actavis)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Riverside Pharmacueticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 190051
Record Dates: First submitted 2019-12-04; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Other

STUDY DESIGN:
Intervention Model Description: * Part I: bioequivalence, food-effect, randomized, open-label, single-dose, 3-period, 6-sequence, crossover design.
  * Part II: multiple-dose (every 4 hours), open-label, 1-period design.
  * Part III: multiple-dose (every 2 hours), open-label, 1-period design. Subjects enrolled in Part II and Part III will be a subset of those who completed Part I.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A (Experimental): 1 x DopaSnap® tablet, administered under fasting conditions.
  Interventions: Drug: DopaSnap®
- Treatment B (Active Comparator): 1 x RLD of CD-LD tablet administered under fasting conditions.
  Interventions: Drug: RDL of CD-LD
- Treatment C (Experimental): Test - fed 1 x DopaSnap® tablet , administered under fed conditions.
  Interventions: Drug: DopaSnap®
- Treatment D (Experimental): DopaSnap® tablet administered at 0 and 4 hours post-first dose, for a total daily dose of CD/LD 50/200 mg.
  Interventions: Drug: DopaSnap®
- Treatment E (Experimental): ½ x DopaSnap® tablet administered at 0, 2, 4, and 6 hours post-first dose
  Interventions: Drug: DopaSnap®

INTERVENTIONS:
Drug: DopaSnap® — immediate release CD/LD 25/100mg; Riverside Pharmaceuticals Corporation, USA
  Other Names: test product
  Arms: Treatment A; Treatment C; Treatment D; Treatment E
Drug: RDL of CD-LD — (immediate release CD/LD 25/100mg; Merck Sharp & Dohme Corp., USA),
  Other Names: Reference
  Arms: Treatment B

SUMMARY:
This will be a single center, bioequivalence and food-effect, open-label study designed to be conducted in three sequential parts:

DETAILED DESCRIPTION:
This will be a single center, bioequivalence and food-effect, open-label study designed to be conducted in three sequential parts:

* Part I: bioequivalence, food-effect, randomized, open-label, single dose, 3-period, 6-sequence, crossover design.
* Part II: multiple-dose (every 4 hours), open-label, 1-period design.
* Part III: multiple-dose (every 2 hours), open-label, 1-period design.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥35 and ≤75 years of age, with BMI > 18.5 and < 30.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing. Subjects vomiting within 24 hours pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Qualified Investigator.
   2. the absence of clinically significant history of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after the last study drug administration:

   1. intra-uterine contraceptive device placed at least 4 weeks prior to study drug administration;
   2. male condom with intravaginally applied spermicide starting at least 21 days prior to study drug administration;
   3. hormonal contraceptives starting at least 4 weeks prior to study drug administration and must agree to use the same hormonal contraceptive throughout the study;
   4. sterile male partner (vasectomized since at least 6 months).
4. Capable of consent.

Exclusion Criteria:

* 1) Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.

  2) Positive urine drug screen, alcohol breath test, or urine cotinine test at screening.

  3) History of allergic reactions to carbidopa, levodopa, or other related drugs, or to any excipient in the formulation.

  4) Positive pregnancy test at screening. 5) Clinically significant ECG abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.

  6) History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).

  7) History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.

  8) Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.

  9) Use of medication other than topical drug products without significant systemic absorption and hormonal contraceptives:
  1. prescription medication within 14 days prior to the first dosing;
  2. over-the-counter products and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 14 days prior to the first dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily);
  3. a depot injection or an implant of any drug within 3 months prior to the first dosing (other than hormonal contraceptives);
  4. MAO inhibitors within 30 days prior to the first dosing; 10) Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.

     11) Hemoglobin < 128 g/L (males) and < 115 g/L (females) and hematocrit < 0.36 L/L (males) and < 0.32 L/L (females) at screening.

     12) Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

     13) Breast-feeding subject. 14) History or presence of myasthenia gravis. 15) Treatment with centrally active drugs or those affecting peripheral cholinergic transmission within 3 months of screening.

     16) The presence of history of narrow angle glaucoma. 17) The presence of history of depression, suicidal tendencies, and other psychotic disorders.

     18) The presence of history of myocardial infarction, arrhythmias, bronchial asthma and other cardiovascular, or pulmonary disease.

     19) The presence of history of melanoma and suspicious undiagnosed skin lesions.

     20) The presence of history of neuroleptic malignant syndrome and non-traumatic rhabdomyolysis.

     21) The presence of history of peptic ulcer disease or undiagnosed recurrent gastro-intestinal bleeding.

     22) The presence of history of convulsions. 23) HAMD-7 score above 3 at screening.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
compare the rate and extent of absorption | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
  • to compare the rate and extent of absorption of the immediate-release CD/LD 25/100 mg DopaSnap® tablet (Test) versus the immediate-release CD-LD tablet (Reference), each administered orally as a single tablet under fasting conditions. AUC0-t
compare the rate and extent of absorption | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
  • to compare the rate and extent of absorption of the immediate-release CD/LD 25/100 mg DopaSnap® tablet (Test) versus the immediate-release CD-LD tablet (Reference), each administered orally as a single tablet under fasting conditions. AUC0-inf
compare the rate and extent of absorption | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
  • to compare the rate and extent of absorption of the immediate-release CD/LD 25/100 mg DopaSnap® tablet (Test) versus the immediate-release CD-LD tablet (Reference), each administered orally as a single tablet under fasting conditions. Cmax
compare the rate and extent of absorption | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
  • to compare the rate and extent of absorption of the immediate-release CD/LD 25/100 mg DopaSnap® tablet (Test) versus the immediate-release CD-LD tablet (Reference), each administered orally as a single tablet under fasting conditions. Residual area
compare the rate and extent of absorption | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
  • to compare the rate and extent of absorption of the immediate-release CD/LD 25/100 mg DopaSnap® tablet (Test) versus the immediate-release CD-LD tablet (Reference), each administered orally as a single tablet under fasting conditions. Tmax
compare the rate and extent of absorption | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
  • to compare the rate and extent of absorption of the immediate-release CD/LD 25/100 mg DopaSnap® tablet (Test) versus the immediate-release CD-LD tablet (Reference), each administered orally as a single tablet under fasting conditions. T½ el
compare the rate and extent of absorption | pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
  • to compare the rate and extent of absorption of the immediate-release CD/LD 25/100 mg DopaSnap® tablet (Test) versus the immediate-release CD-LD tablet (Reference), each administered orally as a single tablet under fasting conditions. Kel
Effect of food on the pharmacokinetics (PK) | A total of 25 blood samples will be collected: pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, and 12 hours post-first dose.
  PK Parameters: AUC0-t
Effect of food on the pharmacokinetics (PK) | A total of 25 blood samples will be collected: pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, and 12 hours post-first dose.
  PK Parameters: Cmax
Effect of food on the pharmacokinetics (PK) | A total of 25 blood samples will be collected: pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, and 12 hours post-first dose.
  PK Parameters: Tmax

SECONDARY OUTCOMES:
PK profile of a fraction of the DopaSnap® tablet | A total of 25 blood samples will be collected: pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, and 12 hours post-first dose.
  • the PK profile of a fraction of the DopaSnap® tablet when administered at frequent intervals every 2 hours comparing to whole tablet every 4 hours PK Parameters: AUC0-t
PK profile of a fraction of the DopaSnap® tablet | A total of 25 blood samples will be collected: pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, and 12 hours post-first dose.
  • the PK profile of a fraction of the DopaSnap® tablet when administered at frequent intervals every 2 hours comparing to whole tablet every 4 hours PK Parameters: Tmax
PK profile of a fraction of the DopaSnap® tablet | A total of 25 blood samples will be collected: pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, and 12 hours post-first dose.
  • the PK profile of a fraction of the DopaSnap® tablet when administered at frequent intervals every 2 hours comparing to whole tablet every 4 hours PK Parameters: Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Lamouche, PhD, Principal Investigator — Syneos Health
Locations (1):
- Syneous Health, Québec, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No